CLINICAL TRIAL: NCT01926496
Title: A Phase 4 Trial Comparing the Cumulative Incidence of SCC After Treatment With Ingenol Mebutate and Imiquimod for Multiple Actinic Keratoses on Face and Scalp. A Multi-centre, Randomised, Two-arm, Open Label, Active-controlled, Parallel Group, 36-month Trial
Brief Title: Risk of Squamous Cell Carcinoma on Skin Areas Treated With Ingenol Mebutate Gel, 0.015% and Imiquimod Cream, 5%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP0041-63; 2012-003112-31 (EudraCT Number)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2020-08

CONDITIONS: Actinic Keratosis (AK)
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ingenol Mebutate (Experimental): Arm A: Ingenol mebutate gel 0.015% applied daily for 3 consecutive days to the selected treatment area followed by 8 weeks' rest. Retreatment for another 3 consecutive days if the treatment field is not completely cleared of AKs at Week 8
  Interventions: Drug: Ingenol Mebutate Gel, 0.015%
- Imiquimod (Active Comparator): Arm B: Imiquimod 5% cream applied 3 days per week for 4 weeks to the selected treatment area followed by 4 weeks' rest. Retreatment for another 4 weeks if the treatment field is not completely cleared of AKs at Week 8
  Interventions: Drug: Imiquimod Cream, 5%

INTERVENTIONS:
Drug: Ingenol Mebutate Gel, 0.015% — Ingenol mebutate gel 0.015 % (Picato®) applied on the selected treatment area. Retreatment if the treatment field is not completely cleared of AKs.
  Other Names: Picato®
  Arms: Ingenol Mebutate
Drug: Imiquimod Cream, 5% — Imiquimod 5% cream applied to the selected treatment area. Retreatment if the treatment field is not completely cleared of AKs
  Other Names: Aldara®
  Arms: Imiquimod

SUMMARY:
The purpose of the study is to compare the risk of developing squamous skin cancer (SCC) or other types of cancer after treatment of AKs with ingenol mebutate gel or imiquimod cream. Subjects will be randomised to treatment with ingenol mebutate or imiquimod and will receive a second treatment cycle with the same treatment if the first treatment does not clear all AKs. Subjects will be followed over a period of three year (36 months) after first treatment

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF) prior to any trial-related procedures
2. Subjects with 5 to 9 clinically typical, visible and discrete AKs within a contiguous 25 cm² treatment area on the face or scalp.
3. Subject at least 18 years of age
4. Female subjects must be of either:

   1. Non-childbearing potential, or,
   2. Childbearing potential, provided there is a confirmed negative urine pregnancy test
5. Female subjects of childbearing potential must be willing to use highly effective methods of contraception (Pearl index < 1%)

Exclusion Criteria:

1. Location of the selected treatment area:

   * on the periorbital skin
   * on the perioral skin/around the nostrils
   * within 5 cm of an incompletely healed wound
   * within 10 cm of a suspected BCC or SCC or other neoplasia
2. Selected treatment area lesions that have atypical clinical appearance (e.g., hypertrophic, hyperkeratotic or cutaneous horn).
3. History of SCC, BCC, malignant melanoma or other neoplasia in the selected treatment area.
4. History or evidence of skin conditions other than the trial indication that would interfere with evaluation of the trial medication in the selected treatment area
5. Use of ingenol mebutate and/or imiquimod in and within 5 cm of the selected treatment area within 2 years prior to Screening (Visit 1)
6. Organ transplant recipients
7. Immunosuppressed subjects (for example HIV patients)
8. Female subjects who are breastfeeding.
9. Subjects who are institutionalised by court order or by the local authority
10. In the opinion of the investigator, the subject is unlikely to comply with the Clinical Study Protocol (e.g. alcoholism, drug dependency or psychotic state)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf-Markus Szeimies, Prof.Dr.med., Principal Investigator — Klinik für Dermatologie und Allergologie
Locations (46):
- France (16):
  - CHU Angers - Service de Dermatologie, Angers
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - HOPITAL AVICENNE - Service de Dermatologie, Bobigny
  - CHRU de Brest - Hôpital Morvan - Service de Dermatologie, Brest
  - CHU Albert Michallon - Service de Dermatologie, Pôle Pluridisciplinaire de Médecine, Grenoble
  - Hôpital Claude Huriez - CHRU de Lille - Clinique de Dermatologie, Lille
  - Hôpital de la Timone - Service de Dermatologie Vénérologie, Marseille
  - CHU de Nantes - Hôtel Dieu - Unité Fonctionnelle de Dermatologie Cancérologie, Nantes
  - HOPITAL DE L ARCHET II - Service de Dermatologie-Vénérologie, Nice
  - Hôpital Caremeau, Nîmes
  - HOPITAL COCHIN TARNIER - Service de Dermatologie, Paris
  - Hôpital Saint Louis - Service de Dermatologie, Paris
  - CHU BORDEAUX - Hôpital Haut-Lévêque, Pessac
  - CHU Poitiers - Service de Dermatologie, Poitiers
  - C.H.U. de Saint-Etienne - Hôpital Nord, Saint-Etienne
  - Hôpital d'instruction des Armées Bégin - Clinique Dermatologique, Saint-Mandé
- Germany (14):
  - Hautarztpraxis Simon, Berlin
  - Hauttumorzentrum Bochum Universitätsklinikum der Ruhr-Universität-Bochum, Bochum
  - Praxis Streit Bucholz, Buchholz
  - Dermatologisches Zentrum, Am Krankenhaus 1, Buxtehude
  - Klinikum Dortmund - Hautklinik, Dortmund
  - Mensingderma, Hamburg
  - Universitätsklinikum Leipzig Klinik für Dermatologie, Venerologie und Allergologie, Leipzig
  - Hautpraxis Dr. Ina Schulze, Markkleeberg
  - Hauttumorzentrum Münster, Münster
  - Klinik für Dermatologie und Allergologie, Klinikum Vest, Behandlungszentrum, Knappschaftskrankenhaus Recklinghausen,, Recklinghausen
  - Universitätklinikum Regensburg, Regensburg
  - Praxis Dr. Hoffmann, Witten
  - Praxis Derma Hübinger, Wuppertal
  - Universitätsklinikum Würzburg, Würzburg
- United Kingdom (16):
  - Ninewells Hospital, Dundee, Angus
  - Cumberland Infirmary, Carlisle, Cumbria
  - Heavitree Hospital, Exeter, Devon
  - Brighton General Hospital, Brighton, East Sussex
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - Monklands Hospital, Airdrie, Lanarkshire
  - Scunthorpe General Hospital, Scunthorpe, Lincolnshire
  - Royal Gwent Hospital, Newport, Monmouthshire
  - Harrogate District Hospital, Harrogate, North Yorkshire
  - Scarborough Hospital, Scarborough, North Yorkshire
  - Cannock Chase Hospital, Cannock, Staffordshire
  - East Surrey Hospital, Redhill, Surrey
  - Southlands Hospital, Shoreham-by-Sea, West Sussex
  - St Luke's Hospital, Bradford, West Yorkshire
  - Chapel Allerton Hospital, Leeds, West Yorkshire
  - Hull Royal Infirmary, Hull

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical trial was performed at 44 sites in 3 countries: France, 11 sites; Germany, 15 sites; and United Kingdom, 18 sites
Groups:
- Ingenol Mebutate: Arm A: Ingenol mebutate gel 0.015% applied daily for 3 consecutive days to the selected treatment area followed by 8 weeks' rest. Retreatment for another 3 consecutive days if the treatment field is not completely cleared of AKs at Week 8>
  > Ingenol Mebutate Gel, 0.015%: Ingenol mebutate gel 0.015 % (Picato®) applied on the selected treatment area. Retreatment if the treatment field is not completely cleared of AKs.
- Imiquimod: Arm B: Imiquimod 5% cream applied 3 days per week for 4 weeks to the selected> treatment area followed by 4 weeks' rest. Retreatment for another 4 weeks if the treatment field is not completely cleared of AKs at Week 8>
  > Imiquimod Cream, 5%: Imiquimod 5% cream applied to the selected treatment area. Retreatment if the treatment field is not completely cleared of AKs
Period: Overall Study
Arm/Group | Ingenol Mebutate | Imiquimod
Started | 240 | 245
Completed | 203 | 197
Not Completed | 37 | 48

BASELINE CHARACTERISTICS:
Population: In total, 485 subjects were randomised (full analysis set), but 1 subject (randomised in United Kingdom) was not treated. To support the primary safety endpoints, all baseline and safety results are based on the 484 subjects. Efficacy analysis are based on all 485 randomized subjects due to the intention-to-treat principle.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ingenol Mebutate | Imiquimod | Total
Number analyzed (Participants) | 240 | 244 | 484
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 42 | 76
  >=65 years | 206 | 202 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (7.1) | 72.0 (8.0) | 72.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 230 | 229 | 459
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 12 | 26
  Not Hispanic or Latino | 226 | 232 | 458
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 240 | 244 | 484
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 80 | 81 | 161
  France | 60 | 63 | 123
  Germany | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Incidence of SCC
Description: Cumulative incidence of SCC after treatment with ingenol mebutate gel and imiquimod cream.> The primary response criterion is diagnosis of SCC (defined as invasive SCC i.e. excludes SCC in situ) in the treatment field across the 3-year trial period.> Kaplan-Meier estimate based on time to SCC or censoring.
Time Frame: 3 years
Population: Safety analysis set: all treated subjects
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Ingenol Mebutate | Imiquimod
Number analyzed (Participants) | 240 | 244
percentage of subjects | 3.1 [1.4 to 6.0] | 0.4 [0.0 to 2.2]

2. Secondary Outcome: Incidence of SCC and Other Neoplasia
Description: Cumulative incidence of SCC and other neoplasia after treatment with ingenol mebutate gel and imiquimod cream.> The secondary response criterion is diagnosis of SCC and other neoplasia in the treatment field across the 3-year trial period.> Kaplan-Meier estimate based on time to SCC and other neoplasia, or censoring.
Time Frame: 3 years
Population: Safety analysis set: all treated subjects
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Ingenol Mebutate | Imiquimod
Number analyzed (Participants) | 240 | 244
percentage of subjects | 6.2 [3.5 to 9.8] | 2.3 [0.9 to 4.9]

3. Secondary Outcome: Number of Participants With Complete Clearance of AK Lesions After Last Treatment
Description: To compare the complete clearance of AK lesions in the selected treatment area after the last treatment cycle (at Week 8 or 16)
Time Frame: 8-16 weeks
Population: Full analysis set: all randomised subjects
Measure: Count of Participants; unit: Participants
Groups:
- Ingenol Mebutate: Arm A: Ingenol mebutate gel 0.015% applied daily for 3 consecutive days to the selected treatment area followed by 8 weeks' rest. Retreatment for another 3 consecutive days if the treatment field is not completely cleared of AKs at Week 8 >
  > Ingenol Mebutate Gel, 0.015%: Ingenol mebutate gel 0.015 % (Picato®) applied on the selected treatment area. Retreatment if the treatment field is not completely cleared of AKs.
- Imiquimod: Arm B: Imiquimod 5% cream applied 3 days per week for 4 weeks to the selected
  > treatment area followed by 4 weeks' rest. Retreatment for another 4 weeks if the treatment field is not completely cleared of AKs at Week 8
  >
  > Imiquimod Cream, 5%: Imiquimod 5% cream applied to the selected treatment area. Retreatment if the treatment field is not completely cleared of AKs
Arm/Group | Ingenol Mebutate | Imiquimod
Number analyzed (Participants) | 240 | 245
Participants | 168 | 192
Statistical Analysis 1: Comparison: Ingenol Mebutate vs Imiquimod; Test type: Superiority; p = 0.03, Cochran-Mantel-Haenszel; Stratified by country, anatomical location and history of squamous cell carcinoma; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.80 to 0.99] — Cochran-Mantel-Haenszel relative risk (ingenol mebutate / imiquimod), stratified by country, anatomical location and history of squamous cell carcinoma

4. Secondary Outcome: Number of Participants With Partial Clearance of AK Lesions
Description: To compare the partial (at least 75%) clearance of AK lesions in the selected treatment area after the last treatment cycle (at Week 8 or 16)
Time Frame: 8-16 weeks
Population: Full analysis set: all randomised subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Ingenol Mebutate | Imiquimod
Number analyzed (Participants) | 240 | 245
Participants | 195 | 210
Statistical Analysis 1: Comparison: Ingenol Mebutate vs Imiquimod; Test type: Superiority; p = 0.18, Cochran-Mantel-Haenszel; Stratified by country, anatomical location and history of squamous cell carcinoma; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.87 to 1.03] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Number of Participants With Complete Clearance of AK Lesions at 12 Months
Description: To compare the complete clearance of AK lesions at 12 months, defined as no AK lesions in the selected treatment area at any time from the last treatment cycle at Week 8 or 16 through to Month 12.
Time Frame: 1 year
Population: Full analysis set: all randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Ingenol Mebutate | Imiquimod
Number analyzed (Participants) | 240 | 245
Participants | 70 | 108
Statistical Analysis 1: Comparison: Ingenol Mebutate vs Imiquimod; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Stratified by country, anatomical location and history of squamous cell carcinoma; Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.52 to 0.84] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: From Day 1 and up to 3 years.
Description: Adverse events (AEs) were reported differently before and after Week 20. Week 20 is the first week of the follow-up period. Before Week 20, all AEs and serious AEs were recorded; after Week 20, all AEs inside the treatment area but only BCC/SCC and related SAEs outside the treatment area, were recorded.
  As per above rules, there were deaths occuring after Week 20 without an associated AE recorded. However, all deaths in the trial are included under "All-Cause Mortality"
Groups:
- Ingenol Mebutate Until Week 20: Ingenol mebutate gel 0.015% applied daily for 3 consecutive days to the selected treatment area followed by 8 weeks' rest. Retreatment for another 3 consecutive days if the treatment field is not completely cleared of AKs at Week 8.
  Ingenol Mebutate Gel, 0.015%: Ingenol mebutate gel 0.015 % (Picato®) applied on the selected treatment area. Retreatment if the treatment field is not completely cleared of AKs.
- Imiquimod Until Week 20: Imiquimod 5% cream applied 3 days per week for 4 weeks to the selected treatment area followed by 4 weeks' rest. Retreatment for another 4 weeks if the treatment field is not completely cleared of AKs at Week 8 Imiquimod Cream, 5%: Imiquimod 5% cream applied to the selected treatment area. Retreatment if the treatment field is not completely cleared of AKs
- Ingenol Mebutate After Week 20: Ingenol mebutate Week 20 is the first week of the follow-up period.
- Imiquimod After Week 20: Imiquimod Week 20 is the first week of the follow-up period.
Arm/Group | Ingenol Mebutate Until Week 20 | Imiquimod Until Week 20 | Ingenol Mebutate After Week 20 | Imiquimod After Week 20
All-Cause Mortality (participants affected / at risk) | 0/240 | 1/244 | 8/240 | 5/244
Serious Adverse Events (participants affected / at risk) | 21/240 | 14/244 | 11/240 | 2/244
Other Adverse Events (participants affected / at risk) | 67/240 | 70/244 | 51/240 | 50/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ingenol Mebutate Until Week 20 (N=240) | Imiquimod Until Week 20 (N=244) | Ingenol Mebutate After Week 20 (N=240) | Imiquimod After Week 20 (N=244)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3) | 2 (2) — Source data does not describe 'number of events', only 'number of subjects'.
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2) | 5 (5) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ingenol Mebutate Until Week 20 (N=240) | Imiquimod Until Week 20 (N=244) | Ingenol Mebutate After Week 20 (N=240) | Imiquimod After Week 20 (N=244)
Eye swelling (Eye disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Application site pain (General disorders) | 22 (28) | 15 (17) | 1 (2) | 0 (0)
Application site pruritus (General disorders) | 14 (15) | 13 (15) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 8 (9) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 16 (19) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (12) | 11 (11) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 12 (15) | 33 (56) | 36 (62)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3) | 24 (42) | 24 (38)
Headache (Nervous system disorders) | 10 (12) | 13 (14) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma seeks publication of all Phase 3 clinical trials in peer-reviewed journals within 18 months of trial completion, regardless of whether the findings are positive or negative. If there is no multi-centre publication within 18 months after the clinical trial has been completed or terminated at all trial sites, the investigator has the right to publish the results from the clinical trial generated by the investigator.

DOCUMENTS (2):
  • Study Protocol (2013-03-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT01926496/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT01926496/SAP_001.pdf